CLINICAL TRIAL: NCT03089684
Title: Correspondence of Dietary Intake and Biomarker Data
Brief Title: Correspondence of Folate Dietary Intake and Biomarker Data
Status: Completed | Type: Observational
Sponsor: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Regan Bailey, Nutritional Epidemiologist, National Institute of Health and Nutrition
Other Study IDs: ODS2015_1
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Folate Deficiency
Keywords: NHANES; Folate; Folic Acid
MeSH Terms: conditions — Folic Acid Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This NHANES analysis compares self-reported dietary folate with serum and red blood cell folate status in U.S. adults.

DETAILED DESCRIPTION:
Background: Public health concerns of both low and high folate status exist in the U.S. Recent publications have questioned the utility of self-reported dietary intake data in research and monitoring.

Objective: The purpose of this analysis was to examine the relationship between self-reported folate intakes and folate status biomarkers, and to evaluate their usefulness for several types of applications.

Design: Usual dietary intakes of folate were examined using the National Cancer Institute (NCI) method to adjust 2, 24-hour dietary recalls (including dietary supplements) for within-person variation and compared these intakes with serum and red blood cell (RBC) folate among 4,878 non-pregnant, non-lactating participants ≥19y in NHANES 2011-2012, a nationally representative, cross-sectional survey, with respect to consistency across prevalence estimates and rank order comparisons.

ELIGIBILITY:
Inclusion Criteria:

* adults, ages 19+ years

Exclusion Criteria:

* missing data
* non-pregnant
* non-lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NHANES is a nationally-representative, cross-sectional study of nutrition and health for individuals residing in the U.S.
Sampling Method: Probability Sample
Enrollment: 4878 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Folate status | Up to 24 months
  Comparison of folate in diet and blood

IPD SHARING:
Plan to Share IPD: Undecided